CLINICAL TRIAL: NCT04923126
Title: SJ901: Phase 1/2 Evaluation of Single Agent Mirdametinib (PD-0325901), a Brain-Penetrant MEK1/2 Inhibitor, for the Treatment of Children, Adolescents, and Young Adults With Low-Grade Glioma
Brief Title: SJ901: Evaluation of Mirdametinib in Children, Adolescents, and Young Adults With Low-Grade Glioma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SJ901; NCI-2021-05912 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2021-05-27; First posted 2021-06-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Low-Grade Glioma; Recurrent Low-Grade Glioma; Progressive Low-Grade Glioma
Keywords: Brain tumors in Adolescent; Brain tumors in Children; Brain tumors in Young Adults; Astrocytic tumor; Glioneuronal tumor; Neuroepithelial tumor, not otherwise specified (NOS); Neuroepithelial tumor, not elsewhere classified (NEC); Pilocytic astrocytoma; Pilomyxoid astrocytoma; Pleomorphic xanthroastrocytoma; Ganglioglioma; Gangliocytoma; Diffuse glioma; Diffuse astrocytoma; Oligodendroglioma; Oligoastrocytoma; Papillary glioneuronal tumor; Rosette-forming glioneuronal tumor; Diffuse leptomeningeal glioneuronal tumor; Central neurocytoma; Extraventricular neurocytoma; Angiocentric glioma; Dysembryoplastic neuroepithelial tumor (DNET); Septal Dysembryoplastic neuroepithelial tumor (DNET); Myxoid glioneuronal tumor; Tectal glioma; Desmoplastic infantile astrocytoma; Desmoplastic infantile ganglioglioma; Polymorphous low-grade neuroepithelial tumor of the young; Multinodular and vacuolating neuronal tumor
MeSH Terms: conditions — Astrocytoma; Neoplasms, Neuroepithelial; Ganglioglioma; Ganglioneuroma; Oligodendroglioma; Neurocytoma | interventions — mirdametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I: Recurrent and/or progressive low-grade glioma without prior exposure to MEK inhibitors (Experimental): Participants will receive mirdametinib at one of the dose levels twice daily days 1-28. For the first cycle of treatment, participants will take mirdametinib tablets dissolved in water. After the first cycle of treatment, participants may receive the medicine the same way (dissolved in water) or may receive capsules. Treatment repeats every 28 days for up to 26 cycles of treatment (24 months) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mirdametinib
- Phase 2, Cohort 1: Newly diagnosed and/or previously untreated (except surgery) (Experimental): Participants will receive the RP2D of mirdametinib. Therapy will be administered in cycles of 28 days and may be continued for up to 24 months (26 cycles) in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mirdametinib
- Phase 2, Cohort 2: Recurrent and/or Progressive without prior exposure to MEK inhibitors (Experimental): Participants will receive the RP2D of mirdametinib. Participants may take mirdametinib tablets dissolved in water, or receive capsules. Therapy will be administered in cycles of 28 days and may be continued for up to 24 months (26 cycles) in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mirdametinib
- Phase 2, Cohort 3a: (Experimental): Participants with recurrent and/or progressive low-grade glioma who previously received ≥ 6 courses MEK inhibitor (including mirdametinib) and did not progress while on active MEKi therapy. Participants will receive the RP2D of mirdametinib. Participants with previous exposure to mirdametinib may receive a starting dose lower than the RP2D, depending on the dose they tolerated during their previous exposure. Participants may take mirdametinib tablets dissolved in water, or receive capsules. Therapy will be administered in cycles of 28 days and may be continued for up to 24 months (26 cycles) in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mirdametinib
- Phase 2, Cohort 3b: (Experimental): Participants with recurrent and/or progressive low-grade glioma who previously received ≥ 6 courses MEK inhibitor (including mirdametinib) and did not progress while on active MEKi therapy. Participants will receive the RP2D of mirdametinib. Participants may take mirdametinib tablets dissolved in water, or receive capsules. Therapy will be administered in cycles of 28 days and may be continued for up to 24 months (26 cycles) in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mirdametinib

INTERVENTIONS:
Drug: Mirdametinib — By mouth, nasogastric (NG) tube or gastrostomy tube (G-tube) BID, days 1-28
  Other Names: PD-0325901

SUMMARY:
This is an open-label, multi-center, Phase 1/2 study of the brain-penetrant MEK inhibitor, mirdametinib (PD-0325901), in patients with pediatric low-grade glioma (pLGG).

DETAILED DESCRIPTION:
The objectives of this study are:

Phase 1

Primary Objectives:

* To determine the safety and tolerability and estimate the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of mirdametinib dosed twice daily on a continuous schedule in pediatric patients with progressive or recurrent low-grade glioma.
* To characterize the plasma pharmacokinetics (PK) of mirdametinib.

Phase 2

Cohort 1: Newly diagnosed and/or previously untreated (except surgery)

Primary Objectives:

* To assess the efficacy, defined as the sustained objective response rate [a Partial Response (PR), Major Response, and/or Complete Response (CR) sustained over 8 weeks] observed over any time on active treatment with mirdametinib in previously untreated patients (except surgery) with WHO grade I or grade II glioma.
* To characterize the plasma pharmacokinetics of mirdametinib in children, adolescents, and young adults with low-grade gliomas.
* To describe the toxicity profile of mirdametinib in pediatric patients.

Secondary Objectives:

* Estimate the efficacy of mirdametinib as measured by progressive free survival (PFS) and overall survival (OS) in patients with previously untreated WHO grade I or grade II glioma.
* To describe treatment responses (Progressive Disease, Stable Disease, Minor Response, Partial Response, Major Response, and Complete Response) observed in previously untreated patients (except surgery) with WHO grade I or grade II glioma over any time on active treatment with mirdametinib.
* To characterize and monitor patient neurocognitive function and quality of life in patients while on study.

Cohort 2: Recurrent and/or Progressive without prior exposure to MEK inhibitors

Primary Objectives:

* To assess the efficacy, defined as the sustained objective response rate (a PR, Major Response, and/or CR sustained over 8 weeks) observed anytime on active treatment with mirdametinib in patients with recurrent and/or progressive WHO grade I or grade II glioma not previously treated with MEK inhibitors.
* To characterize the plasma pharmacokinetics of mirdametinib in children, adolescents, and young adults with low-grade gliomas.
* To describe the toxicity profile of mirdametinib in pediatric patients with recurrent or progressive disease, not previously treated with MEK inhibitors.

Secondary Objectives:

* Estimate the efficacy of mirdametinib as measured by PFS and OS in patients with recurrent and/or progressive WHO grade I or grade II glioma not previously treated with MEKi
* To describe treatment responses (Progressive Disease, Stable Disease, Minor Response, Partial Response, Major Response, and Complete Response) observed in patients with recurrent and/or progressive WHO grade I or grade II glioma without prior exposure to MEK inhibitors.
* To characterize and monitor patient neurocognitive function and quality of life in patients while on study.

Cohort 3: Re-treatment (recurrent and/or progressive disease previously treated with a MEK inhibitor)

Primary Objectives:

* To estimate the 1-year disease stabilization rate (defined as lack of disease progression for ≥ 12 courses of mirdametinib) in patients with recurrent and/or progressive WHO grade I or grade II glioma who previously received ≥ 6 courses MEK inhibitor (including mirdametinib) and did not progress while on active MEKi therapy (cohort 3A).
* To estimate the 6-month disease stabilization rate (defined as lack of disease progression for ≥ 6 courses of mirdametinib) in patients with recurrent and/or progressive WHO grade I or grade II glioma who previously received a MEK inhibitor, other than mirdametinib, and progressed while on active MEKi therapy (cohort 3B).
* To characterize the plasma pharmacokinetics of mirdametinib in children, adolescents, and young adults with low-grade gliomas.
* To describe the toxicity profile of mirdametinib in pediatric patients with recurrent or progressive disease, previously treated with MEK inhibitors.

Secondary Objectives:

* Estimate the efficacy of mirdametinib as measured by PFS and OS in patients with recurrent and/or progressive WHO grade I or grade II glioma previously treated with MEK inhibitors
* To describe treatment responses (Progressive Disease, Stable Disease, Minor Response, Partial Response, Major Response, and Complete Response) observed in patients with recurrent and/or progressive WHO grade I or grade II glioma previously treated with a MEK inhibitor.
* To characterize and monitor patient neurocognitive function and quality of life in patients while on study.

SJ901 will proceed in two phases. Phase 1 will evaluate the safety, tolerability and pharmacokinetics of mirdametinib when dosed continuously up to 3 mg/m^2/dose twice daily (BID) in patients with progressive or recurrent pLGG without prior MEK inhibitor (MEKi) exposure. This phase will identify the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) and will contain a small expansion cohort before launching phase 2. Phase 2 will utilize the MTD/RP2D to evaluate mirdametinib efficacy, pharmacokinetics, safety and tolerability in broader cohorts of patients with newly diagnosed or progressive/recurrent pLGG (+/- prior MEK inhibitor exposure).

In Phase 1 of the study, participants with progressive or recurrent pLGG without prior MEKi exposure are eligible and will be enrolled onto a single dose level. The Rolling 6 design will be used to estimate the MTD/RP2D and to determine the dose limiting toxicities (DLTs) of the escalating doses. Once a candidate MTD or RP2D based on 6 subjects has been determined additional evaluable subjects will be enrolled as part of a Phase 1 expansion cohort in order to better describe the safety and tolerability of the MTD/RP2D. The data from all subjects treated at the MTD/RP2D (patients from the dose-finding/dose-escalation study plus expansion cohort) will also be used to assess the stage I efficacy criteria for cohort 2 as part of the Phase 2 design. If these criteria are met, cohort 2 sample size will be expanded beyond the interim analysis and the Phase 2 study will be initiated in cohort 1.

Mirdametinib will be administered twice daily in cycles of 28 days and may be continued for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity. Doses will be based on the BSA calculated before each cycle of therapy. During the DLT period (i.e., cycle 1), all phase 1 participants (including those in the phase 1 expansion cohort) will receive mirdametinib in dispersible tablets only. Thereafter, patients who can swallow capsules may transition to capsules if permitted by their specific dose level.

Once the phase 2 is open to enrollment, participants from the phase 1 on a dose level that differs from the RP2D, may choose to change to the RP2D as long as they have not undergone a dose-reduction for toxicity, and if the treating physician and the patient/family agree it is in the best interest of the patient.

In Phase 2 of the study, participants will be stratified into 3 disease cohorts:

* Cohort 1: Patients with Newly Diagnosed Low-Grade Glioma
* Cohort 2: Patients with Progressive or Recurrent Low-Grade Glioma without Previous MEKi Exposure
* Cohort 3: Patients with Progressive or Recurrent Low-Grade Glioma with Previous MEKi Exposure and:

  * Cohort 3A: Previously received 6 or more cycles of MEKi therapy and did not progress on MEKi therapy
  * Cohort 3B: Previously treated with MEKi, other than mirdametinib, and progressed while on MEKi therapy

Therapy will be administered at RP2D in cycles of 28 days and may be continued for up to 24 months (26 cycles) in absence of disease progression or unacceptable toxicity. Patients in Cohort 3 with previous exposure to mirdametinib may receive a starting dose lower than the RP2D, depending on the dose they tolerated during their previous exposure. For patients enrolled prior to Amendment 4 activation, we will utilize dispersible tablet formulation of the study drug. For patients who are enrolled after Amendment 4 activation, we will utilize both the dispersible tablet and capsule formulations.

ELIGIBILITY:
Inclusion Criteria: Screening Phase

* Participants with histologically confirmed or suspected low-grade glioma, including neuronal and mixed neuronal-glial tumors
* Participant must have adequate tumor tissue from primary and/or relapsed tumor for central pathology review
* For Phase 1: Projected to be ≥ 2 years and < 25 years at the time of study enrollment
* Participant's body surface area (BSA) at time of study enrollment must fall within the range outlined in the protocol for the specific dose level under evaluation:

  * Phase 1: Dose Finding/Dose-escalation

    * For Phase 1 participant's BSA must fall within the range specified in the protocol for the specific dose level under evaluation.
  * Phase 2: All Cohorts:

    * For Phase 2 of the study the upper BSA restrictions will be removed.
* Participant and/or guardian can understand and is willing to sign a written informed consent document according to institutional guidelines

Exclusion Criteria: Screening Phase

* Participants with known current retinal pathology that is consistent with or a precursor for central serous retinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration
* Participants with a known malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of mirdametinib (e.g., gastric bypass, lap band, or other gastric procedures)
* Participant with a known history of liver disease or known hepatic or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones)
* Participants with a clinically significant history of chronic interstitial lung disease (such as bronchopulmonary dysplasia, chronic bronchiolitis, obliterative bronchiolitis, chronic aspiration pneumonia, surfactant protein disorder, or other serious chronic pulmonary condition). Participants with a history of asthma, reactive airways disease, or viral pneumonitis are not to be excluded if disease has resolved or is well-controlled.

Inclusion Criteria: Phase 1 and Phase 2, All Cohorts

* Participant must be ≥ 2 years and < 25 years of age at the time of enrollment
* Participant's BSA at time of study enrollment must fall within the range outlined below for the specific dose level under evaluation:

  * Phase 1: Dose-finding/Dose-escalation

    * For Phase 1 participant's BSA must fall within the range specified in the protocol for the specific dose level under evaluation.
  * Phase 2: All Cohorts

    * For Phase 2 of the study the upper BSA restrictions will be removed.
* Participant must have confirmation of one of the following diagnosis per St. Jude Children's Research Hospital central pathology review of primary and/or relapsed tumor:

  * Eligible tumors include:

    * Low-grade glioma/astrocytic tumor/glioneuronal tumor/neuroepithelial tumor, not otherwise specified (NOS) or not elsewhere classified (NEC)
    * Pilocytic astrocytoma
    * Pilomyxoid astrocytoma
    * Pleomorphic xanthroastrocytoma
    * Ganglioglioma
    * Gangliocytoma
    * Diffuse glioma, diffuse astrocytoma, oligodendroglioma, or oligoastrocytoma
    * Papillary glioneuronal tumor
    * Rosette-forming glioneuronal tumor
    * Diffuse leptomeningeal glioneuronal tumor
    * Central neurocytoma, extraventricular neurocytoma
    * Angiocentric glioma
    * Dysembryoplastic neuroepithelial tumor (DNET), septal DNET, myxoid glioneuronal tumor
    * Tectal glioma
    * Desmoplastic infantile astrocytoma / ganglioglioma
    * Polymorphous low-grade neuroepithelial tumor of the young
    * Multinodular and vacuolating neuronal tumor
* In addition, tumor on central review must show evidence supporting MAPK pathway activation as defined by IHC, FISH and/or DNA/RNA sequencing (i.e. BRAF fused or rearranged, FGFR1/2/3 aberration, NF1, NF2, PTPN11, SOS1, RAF1 mutations, MYB or MYBL1 fused or rearranged, etc.) or occur in a participant with known NF1, NF2, SOS1, RAF1, or PTPN11 germline mutation. (Note: tests that show evidence supporting MAPK pathway activation that have been already performed do not need to be repeated as long as deemed acceptable by central review).
* Participant must have measurable or evaluable disease (as defined in the protocol)

  * Note: Participants with metastatic disease or multiple independent primary LGGs are allowed on study.
* Participants who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to enrollment with no plans for escalation.
* Participant must have a Lansky (<16 years) or Karnofsky (≥16 years) performance score of ≥ 50 and, in the opinion of the investigator, a minimum life expectancy of at least 6 weeks.

  * Note: Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Participant must have adequate bone marrow and organ function as defined as:

  * ANC ≥ 1.0 x 10^9/L without growth factor support within 7 days
  * Platelet count ≥ 75x 10^9/L without support of a platelet transfusion within 7 days
  * Hemoglobin ≥8.0 g/dL without support of a blood transfusion within 7 days
  * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus must be ≤ grade 1 or corrected to ≤ grade 1 with supplements before first dose of study medication
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN. For the purposes of this study the ULN of ALT and AST is 45 U/L.
  * Total bilirubin ≤ ULN; or if > ULN then direct bilirubin ≤ 1.5 x ULN
* Adequate renal function defined as:

  * Serum creatinine ≤ the maximum serum creatinine based on age/gender: Age: 2 to < 6 years: maximum serum creatinine (mg/dL) 0.8 (male, female), Age: 6 to <10 years: maximum serum creatinine (mg/dL) 1 (male, female), Age: 10 to <13 years: maximum serum creatinine (mg/dL) 1.2 (male, female), Age: 13 to <16 years: maximum serum creatinine (mg/dL) 1.5 (male); 1.4 (female), Age: ≥ 16 years: maximum serum creatinine (mg/dL) 1.7 (male); 1.4 (female)
* Adequate cardiac function defined as:

  * LVEF > 50% by ECHO
  * QTc interval ≤ 450 msec for male participants, ≤ 470 msec for female participants after electrolytes have been corrected.
* Hypertension:

  * Patients 2-12.99 years of age must have a blood pressure that is ≤ 95th percentile +10 mmHg for age, height, and gender at the time of enrollment (with or without the use of anti-hypertensive medications).
  * Patients ≥ 13 years of age must have a blood pressure ≤ 140/90 mmHg at the time of enrollment (with or without the use of anti-hypertensive medications).

    * Note for patients of all ages: Adequate blood pressure can be achieved using medication for the treatment of hypertension.
* Participants of childbearing/child-fathering potential must agree to use contraception.
* Participants and/or guardian have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.
* Participants who are receiving P-gp and BCRP inhibitors must have received their last dose a week or 5 half-lives (whichever is greater) prior to the first mirdametinib dose.

Inclusion Criteria: Phase 1: Progressive or Recurrent Low-Grade Glioma without Previous MEKi exposure

* Participant's tumor must have unambiguously progressed, relapsed, or recurred during or after the most recent prior therapy (chemotherapy or radiotherapy) and pseudoprogression or treatment-related tumor changes have, in the opinion of the investigator, been thoroughly vetted.

  * Progression may be radiographic or clinical (i.e. vision deterioration thought to be related to tumor in patients with optic pathway tumors, or neurologic deterioration thought to be related to tumor) but it must be unequivocal and sufficient to warrant treatment in the opinion of the investigator.
* Prior therapy:

  * Patients who have received the following:

    * ≤ 3 prior treatment regimens with either myelosuppressive chemotherapy or biologic agents and/or
    * focal radiotherapy
* Note that a treatment regimen is defined as a single agent (chemotherapeutic or biologic), or a sequential combination of therapies that can include radiotherapy (with or without concurrent radiosensitizer, chemotherapy, or biologic therapy) followed by maintenance therapy (either single or combination) given over a period of time at either diagnosis or relapse.
* Chemotherapy:

  * Participant must have received their last dose of myelosuppressive anticancer chemotherapy at least 21 days prior to study enrollment or at least 42 days if nitrosourea.
* Monoclonal antibody treatment and agents with known prolonged half-lives:

  * Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment
* MEK inhibitors:

  * Patients must not have received prior exposure to any MEK inhibitors
* XRT/External Beam Irradiation including Protons:

  * Participant must have had their last fraction of radiation ≥ 3 months prior to study enrollment

Inclusion Criteria: Phase 2, Cohort 1: Newly Diagnosed and/or previously untreated (except surgery) Low-Grade Glioma

* No prior anti-cancer treatment except surgery.
* In the opinion of the investigator tumor must warrant treatment defined as any of the following: unsafe to observe, unequivocally progressing on serial imaging, tumor is causing or at high risk of causing neurologic or vision-related deficits.

Inclusion Criteria: Phase 2, Cohort 2: Progressive or Recurrent Low-Grade Glioma without Previous MEK Inhibitor Exposure

* Participant's tumor must have unambiguously progressed, relapsed, or recurred during or after the most recent prior therapy (chemotherapy or radiotherapy) and pseudoprogression or treatment-related tumor changes have, in the opinion of the investigator, been thoroughly vetted.

  * Progression may be radiographic or clinical (i.e. vision deterioration thought to be related to tumor in patients with optic pathway tumors, or neurologic deterioration thought to be related to tumor) but it must be unequivocal and sufficient to warrant treatment in the opinion of the investigator.
* Prior therapy:

  * Chemotherapy:

    * Participant must have received their last dose of myelosuppressive anticancer chemotherapy at least 21 days prior to study enrollment or at least 42 days if nitrosourea.
  * Monoclonal antibody treatment and agents with known prolonged half-lives:

    * Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment
  * MEK inhibitors:

    * Patients must not have received prior exposure to any MEK inhibitors
  * XRT/External Beam Irradiation including Protons:

    * Participant must have had their last fraction of radiation ≥ 3 months prior to study enrollment.
* Note that for this cohort, there are no limitations on number of prior treatment regimens and participants who have received craniospinal radiation are eligible

Inclusion Criteria: Phase 2, Cohort 3: Progressive or Recurrent Low-Grade Glioma with Previous MEK inhibitor Exposure

* Cohort 3A (MEKi responders): Patients who previously received 6 or more cycles of any MEK inhibitor (including mirdametinib) and did NOT progress while on active MEK inhibitor therapy.

  * The progression must have occurred off MEK inhibitor therapy
  * Participant's tumor must have unambiguously relapsed or clinically progressed. Progression may be radiographic or clinical (i.e. vision deterioration thought to be related to tumor in patients with optic pathway tumors, or neurologic deterioration thought to be related to tumor) but it must be unequivocal and sufficient to warrant treatment in the opinion of the investigator.
  * Patient must not have discontinued MEKi (specifically mirdametinib) for unacceptable toxicity, and in the opinion of the PI be able to tolerate subsequent courses of MEKi therapy.
  * Patients must have received treatment with a MEK inhibitor for ≥6 cycles and showed no signs of progression while on active MEK inhibitor therapy.
  * Patients who received additional anti-tumor therapy following discontinuation of MEK inhibitor can be enrolled in this cohort.
* Prior Therapy:

  * Chemotherapy:

    * Participant must have received their last dose of myelosuppressive anticancer chemotherapy at least 21 days prior to study enrollment or at least 42 days if nitrosourea.
  * Monoclonal antibody treatment and agents with known prolonged half-lives:

    * Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment.
  * MEK inhibitors:

    * Participant must have received their last dose of MEKi at least 3 weeks prior to study enrollment.
  * XRT/External Beam Irradiation including Protons:

    * Participant must have had their last fraction of radiation ≥ 3 months prior to study enrollment.
* Note that for this cohort, there are no limitations on number of prior treatment regimens and participants who have received craniospinal radiation are eligible
* Cohort 3B (MEKi non-responders): Patients with previous exposure to alternative MEK inhibitors (excluding mirdametinib) who progressed while on active MEK inhibitor therapy

  * Participant's tumor must have unambiguously relapsed or clinically progressed.
  * Progression may be radiographic or clinical (i.e. vision deterioration thought to be related to tumor in patients with optic pathway tumors, or neurologic deterioration thought to be related to tumor) but it must be unequivocal and sufficient to warrant treatment in the opinion of the investigator. Progression or recurrence must have occurred while on active MEK inhibitor therapy (excluding mirdametinib)
  * Participants are eligible regardless of how many prior cycles were received or prior history of response (i.e. PR, Major Response, or CR)
* Patients who received additional anti-tumor therapy following discontinuation of MEK inhibitor can be enrolled in this cohort as long as they meet the above criteria.
* Prior Therapy:

  * Chemotherapy:

    * Participant must have received their last dose of myelosuppressive anticancer chemotherapy at least 21 days prior to study enrollment or at least 42 days if nitrosourea.
  * Monoclonal antibody treatment and agents with known prolonged half-lives:

    * Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment.
  * Alternative MEK inhibitor:

    * Participant must have received their last dose of MEKi (excluding mirdametinib) at least 3 weeks prior to study enrollment.
  * XRT/External Beam Irradiation including Protons:

    * Participant must have had their last fraction of radiation ≥ 3 months prior to study enrollment.
* Note that for this cohort, there are no limitations on number of prior treatment regimens and participants who have received craniospinal radiation are eligible.

Exclusion Criteria: Phase 1 and Phase 2, All Cohorts

* Participants whose tumor on central review is any of the following:

  * High-grade (WHO III or IV)
  * Subependymal giant cell astrocytoma
  * Ependymoma
  * Histone H3 K27M/K28M or G34/G35-mutant
  * BRAF V600 mutant
  * NTRK1/2/3, ALK, or ROS1 fusion-positive
  * IDH 1/2 mutant
* Participant who is currently receiving any other anticancer or investigational agents (^11C-methionine allowed) or still recovering from acute toxicity potentially related to the agent.
* Ophthalmologic Conditions

  * Patients with central serous retinopathy
  * Patients with retinal vein occlusion or retinal detachment
  * Patients with uncontrolled glaucoma

    * If checking pressure is clinically indicated and feasible per patient's age and ability to complete exam, patients with IOP > 22 mmHg or ULN adjusted by age are not eligible
* Participants with other clinically significant medical disorders (i.e. serious infections or significant cardiac, pulmonary, hepatic, psychiatric, or other organ dysfunction) that in the investigator's judgement could compromise their ability to tolerate or absorb protocol therapy or would interfere with the study procedures or results.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 16 weeks after stopping study therapy are not eligible.
* Participants are excluded if unable to comply with protocol guidelines.

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Estimate the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of mirdametinib dosed twice daily on a continuous schedule in pediatric patients with progressive or recurrent low-grade glioma. | 1 month after start of mirdametinib treatment
  The maximum tolerated dose (MTD) is empirically defined as the highest dose level at which six patients have been treated with at most one patient experiencing a dose-limiting toxicity (DLT) and the next higher dose level determined to be too toxic. The MTD estimate will not be available if the lowest dose level studied is too toxic or the highest dose level studied is considered safe. In the latter case, the highest studied safe dose may be considered as the recommended phase 2 dose (RP2D). The MTD estimation will be limited to evaluable patients and toxicity assessments from course 1 (28 days). We will require that at least 12 DLT evaluable subjects are assessed before the MTD/RP2D is declared.
Phase 1: Determine the safety and tolerability of mirdametinib dosed twice daily on a continuous schedule in pediatric patients with progressive or recurrent low-grade glioma. | Up to 25 months after start of mirdametinib treatment
  Incidence of adverse event data at least possibly related to treatment will be summarized in cohort specific tables by grade and attribution throughout treatment.
Characterize the maximum plasma concentration and area under the concentration-time curve (AUC0-8h) of mirdametinib. | Course 1: Days 1 and 15
  Mirdametinib plasma concentration will be provided and area under the curve (AUC0-8h) estimated based on course 1, days 1 and 15 PK samples
Phase 2, Cohort 1: Objective response rate observed anytime during active treatment and sustained for at least 8 weeks | Up to 24 months after start of mirdametinib treatment
  The response rate, defined as the rate of minor response, partial response (PR), major response, or complete response (CR) will be calculated as the percentage of confirmed responders among all response assessable patients. These rates as well as their exact confidence intervals will be provided and will be summarized by each response category (i.e., PR, major response, and CR). Subjects without an assessment will be considered non-responders.
Phase 2, Cohort 2: Objective response rate observed anytime during active treatment and sustained for at least 8 weeks | Up to 24 months after start of mirdametinib treatment
  The response rate, defined as the rate of minor response, partial response (PR), major response, or complete response (CR) will be calculated as the percentage of confirmed responders among all response assessable patients. These rates as well as their exact confidence intervals will be provided and will be summarized by each response category (i.e., PR, major response, and CR). Subjects without an assessment will be considered non-responders.
Phase 2, Cohort 3a: Estimate 1-year disease stabilization rate | Up to 12 months (slight departures from this timing allowed based on MRI screening) after start of mirdamentinib treatment
  Rate of stable disease from start of treatment until the time of progression or time of last follow-up.
Phase 2, Cohort 3b: Estimate 6-month disease stabilization rate | Up to 6 months (slight departures from this timing allowed based on MRI screening) after start of mirdametinib treatment
  Rate of stable disease from start of treatment until the time of progression or time of last follow-up.
Describe the toxicity profile of mirdametinib by cohort. | Up to 25 months after start of mirdametinib treatment
  Incidence of adverse event data at least possibly related to treatment will be summarized in cohort specific tables by grade and attribution throughout treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) by cohort | Up to 5 years after the last enrolled patient starts treatment
  PFS will be measured using Kaplan Meier approaches from the date of initial treatment to the earliest date of progressive disease, death due to any cause, or date last follow-up.
Rates of Minor Response, by cohort | Up to 5 years after the last enrolled patient starts treatment
  Minor Response is defined as a 25-49% reduction in target lesion area relative to baseline measurements. Overall, the patient should be clinically stable or have improved on physical examination and functional or neurological assessment. Responses and duration will be measured for each cohort from the date of initial treatment to the earliest date of progressive disease, or data of last follow-up.
Rates of Partial Response (PR), by cohort | Up to 5 years after the last enrolled patient starts treatment
  Partial Response (PR) is defined as a 50-75% reduction in the target lesion area relative to baseline measurements. Overall, the patient should be clinically stable or have improved on physical examination and functional or neurological assessment. Responses and duration will be measured for each cohort from the date of initial treatment to the earliest date of progressive disease, or data of last follow-up.
Rates of Major Response, by cohort | Up to 5 years after the last enrolled patient starts treatment
  Major Response is defined as more than 75% reduction in target lesion area relative to baseline measurements. Overall, the patient should be clinically stable or have improved on physical examination and functional or neurological assessment. Responses and duration will be measured for each cohort from the date of initial treatment to the earliest date of progressive disease, or data of last follow-up.
Rates of Complete Response (CR), by cohort | Up to 5 years after the last enrolled patient starts treatment
  Complete Response is defined as disappearance of the target lesion and, if applicable, all areas of metastatic disease as compared to reference scan (baseline or best recorded MRI). Overall, the patient should be clinically stable or have improved on physical examination and functional or neurological assessment. Responses and duration will be measured for each cohort from the date of initial treatment to the earliest date of progressive disease, or data of last follow-up.
Rates of Stable Disease, by cohort | Up to 5 years after the last enrolled patient starts treatment
  Stable disease is defined as an increase or decrease in target lesion area that is not sufficient to qualify as progressive or responsive disease (i.e. minor, partial, major, or complete). Overall, the patient should be clinically stable or have improved on physical examination and functional or neurological assessment. Responses and duration will be measured for each cohort from the date of initial treatment to the earliest date of progressive disease, or data of last follow-up.
Rates of Progressive Disease (PD), by cohort | Up to 5 years after the last enrolled patient starts treatment
  Progressive Disease is defined as any of the following: A greater than 25% increase in target lesion area relative to reference scan, the development of a new tumor lesion, substantial growth (>25%) of a measurable metastatic lesion, or worsening of clinical and/or functional assessment directly related to tumor progression. Responses will be measured for each cohort from the date of initial treatment to the earliest date of progressive disease, or data of last follow-up.
Longitudinal change in intellectual function, by cohort | Baseline (at enrollment), 9 months, 2 years, and 5 years after start of mirdametinib treatment
  To evaluate the effects of mirdametinib treatment on intellectual function among children treated for low-grade glioma. This will be assessed in children 2.6-5.11 years of age using Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV), in children 6-16.11 years of age using the Wechsler Intelligence Scale for Children (WISC-V), and for children 17 years and older using Wechsler Adult Intelligence Scale (WAIS-IV). Scores for each measure will be summarized by timepoint and cohort using descriptive statistics and appropriate plots.
Longitudinal change in attention and executive functions, by cohort | Baseline (at enrollment), 6 months, 9 months, 2 years, 3 years, 4 years, and 5 years after start of mirdametinib treatment
  To evaluate the effects of mirdametinib treatment on attention and executive function in children treated for low-grade glioma. This will be assessed using different instruments as age appropriate: Cogstate will be used to measure attention, working memory and processing speed in children 4 years and older; WPPSI-IV (4-5.11 years of age), WISC-V (6-16.11 years of age) and WAIS-IV (17 years of age and older) will assess brief attention and working memory; Kaufman Test of Educational Achievement, Third Edition (KTEA-3) will assess verbal fluency in children 4-25 years of age; and Behavior Rating Inventory of Executive Function (BRIEF; BRIEF-2) will assess behavioral manifestations of executive function. Scores for each measure will be summarized by timepoint and cohort using descriptive statistics and appropriate plots.
Longitudinal change in memory, by cohort | 9 months, 2 years, and 5 years after start of mirdametinib treatment
  To evaluate the effects of mirdametinib treatment on memory in children treated for low-grade glioma. This will be assessed using different instruments as age appropriate: California Verbal Learning Test, Children's Version (CVLT-C) will be used to measure verbal list learning in children 6-16.11 years of age; the NEPSY-II Memory for Designs subtest (ages 6-16.11) and Wechsler Memory Scale (WMS-IV, ages 17 and older ) will assess nonverbal memory; the Children's Memory Scale (CMS, ages 5-16.11) and WMS-IV (ages 17 and older) Story Memory subtests will assess immediate recall, delayed recall, and recognition of details. Scores for each measure will be summarized by timepoint and cohort using descriptive statistics and appropriate plots.
Longitudinal change in processing speed, by cohort | 9 months, 2 years, and 5 years after start of mirdametinib treatment
  To evaluate the effects of mirdametinib treatment on processing speed in children treated for low-grade glioma. This will be assessed using the age appropriate Wechsler Processing Speed Index [WPPSI-IV (ages 4-5.11), WISC-V (ages 6-16), and WAIS-IV (ages 17 and older)]. Scores for each measure will be summarized by timepoint and cohort using descriptive statistics and appropriate plots.
Longitudinal change in academic achievement, by cohort | 2 years and 5 years after start of mirdametinib treatment
  To evaluate the effects of mirdametinib treatment on academic achievement in children treated for low-grade glioma. Reading and math abilities will be assessed using age-appropriate KTEA-3 subtests: Letter & Word Recognition (ages 4 and older), Word Recognition Fluency (ages 6 and older), Math Computation (ages 5 and older), and Math Fluency (ages 6 and older). Scores for each measure will be summarized by timepoint and cohort using descriptive statistics and appropriate plots.
Longitudinal change in psychosocial functioning, by cohort | Baseline (at enrollment), 6 months, 9 months, 2 years, 3 years, 4 years, and 5 years after start of mirdametinib treatment
  To evaluate the effects of mirdametinib treatment on psychosocial function in children treated for low-grade glioma. Social-emotional measures will include the Behavior Assessment System for Children, Third Edition (BASC-3, ages 2-20.11) to assess behavioral, emotional, and adaptive functioning, as well as the PedsQL (ages 2 and older) to assess health-related quality of life. Scores for each measure will be summarized by timepoint and cohort using descriptive statistics and appropriate plots.
Longitudinal change in adaptive behavior, by cohort | Baseline (at enrollment), 9 months, 2 years, and 5 years after start of mirdametinib treatment
  To evaluate the effects of mirdametinib treatment on adaptive behavior in children treated for low-grade glioma. This will be assessed using the Adaptive Behavior Assessment System, Third Edition (ABAS-3, ages 2-21.11), which rates the child's ability to independently perform age-appropriate daily living skills. Scores will be summarized by timepoint and cohort using descriptive statistics and appropriate plots.

CONTACTS AND LOCATIONS:
Overall Officials: Giles W. Robinson, MD, Principal Investigator — St. Jude Children's Research Hospital; Anna Vinitsky, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — http://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042...